CLINICAL TRIAL: NCT04551131
Title: Use Of A Response-Adapted Ruxolitinib-Containing Regimen For The Treatment Of Hemophagocytic Lymphohistiocytosis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Incyte Corporation (Industry); North American Consortium for Histiocytosis (Other); Cures Within Reach (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLHRUXO; NCI-2020-08320 (Registry Identifier: NCI Clinical Trial Registration)
Record Dates: First submitted 2020-09-02; First posted 2020-09-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Hemophagocytic lymphohistiocytosis; Newly Diagnosed; Frontline therapy; Refractory; Relapsed; Response-adapted; Salvage therapy
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Recurrence | interventions — ruxolitinib; Dexamethasone; Calcium Dobesilate; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Frontline Arm (Experimental): Safety Phase:
  Patients with newly diagnosed HLH will receive ruxolitinib PO or NGT and dexamethasone, PO or IV. Etoposide IV will be added based on disease response.
  Expansion Phase:
  Patients with newly diagnosed HLH treatment will begin with ruxolitinib PO or NGT at the MTD dose. Dexamethasone will be administered PO or IV. Etoposide IV will be added based on disease response.
  Interventions: Drug: Ruxolitinib; Drug: Dexamethasone; Drug: Etoposide
- Salvage Arm (Experimental): Patients with relapsed/refractory HLH will receive ruxolitinib PO or NGT and dexamethasone PO or IV. Etoposide IV will be added based on disease response.
  Interventions: Drug: Ruxolitinib; Drug: Dexamethasone; Drug: Etoposide

INTERVENTIONS:
Drug: Ruxolitinib — Given orally (PO) or per nasogastric tube (NGT) twice a day for 8 weeks
  Other Names: Jakafi®
Drug: Dexamethasone — Given intravenously (IV) or orally (PO) twice a day for 8 weeks
  Other Names: Decadron®; Hexadrol®; Dexone®; Dexameth®
Drug: Etoposide — Given intravenously (IV) once a week for 8 weeks
  Other Names: Etoposide Phosphate; VePesid®; Etopophos®; VP-16

SUMMARY:
This study is a multi-site Phase Ib/II, 2-arm non-randomized clinical trial to determine the efficacy and tolerability of a response-adapted regimen combining ruxolitinib, dexamethasone, and etoposide as Frontline therapy for patients with newly diagnosed hemophagocytic lymphohistiocytosis (HLH) or as Salvage therapy for patients with relapsed/refractory HLH.

Primary Objective

* To determine the efficacy and tolerability of a response-adapted ruxolitinib-containing regimen for patients with newly diagnosed HLH.

Secondary Objectives

* To describe the efficacy and tolerability of a response-adapted ruxolitinib-containing regimen for patients with relapsed/refractory HLH.
* To describe the overall response and outcome for patients with newly diagnosed or relapsed/refractory HLH who are treated with this response-adapted ruxolitinib-containing regimen.

Exploratory Objectives

* To estimate the pharmacokinetic (PK) parameters of ruxolitinib, assess covariates of ruxolitinib pharmacokinetics, and test whether the drug's effectiveness is correlated with systemic drug exposure.
* To query specific immunologic biomarkers and determine whether the levels of these biomarkers correlate with disease response and outcome.

DETAILED DESCRIPTION:
Frontline Arm: Safety Phase and Expansion Phase

Safety Phase: The Frontline Arm will begin with a Safety Phase to identify a feasible and safe dose of ruxolitinib to be given in combination with the "gold standard" HLH-directed agents dexamethasone and etoposide using a response-adapted approach. For this part of the trial, a minimum of 6 newly diagnosed HLH patients will be included. These patients will first receive ruxolitinib 25 mg/m^2/dose by mouth BID (twice a day) and dexamethasone 5 mg/m^2/dose PO or IV BID. For patients whose HLH responds favorably (as outlined in the protocol), ruxolitinib will be continued for 8 weeks if it is tolerated. Dexamethasone will be weaned, as tolerated, over 8 weeks and then discontinued. For patients whose HLH does not respond favorably (as outlined in the protocol), etoposide 150 mg/m2 IV weekly will be added. The dose of ruxolitinib may be escalated or de-escalated as needed, based on observed toxicities and surrogates of disease response.

Expansion Phase: When a dose of ruxolitinib deemed feasible and safe is identified, the Expansion Phase of the Frontline Arm will begin. Patients with newly diagnosed HLH in the Expansion Phase will receive ruxolitinib (at the maximally tolerated dose [MTD] established in the Safety Phase) and dexamethasone 5 mg/m^2/dose by mouth or IV BID. For patients whose HLH responds favorably (as outlined in the protocol), ruxolitinib will be continued for 8 weeks if it is tolerated. Dexamethasone will be weaned, as tolerated, over 8 weeks and then discontinued. For patients whose HLH does not respond favorably (as outlined in the protocol), etoposide 150 mg/m^2 IV weekly will be added. The first dose of dexamethasone will be given at least 8 hours after the first dose of ruxolitinib for PK testing purposes, but patients will not be excluded if dexamethasone has already been started before initiating of ruxolitinib. Disease response evaluations will be completed at 1, 2, 4, 6, and 8 weeks. Treatment will be individualized based on response.

Patients whose HLH responds favorably after 1 week (SD 8) of therapy (e.g., favorable response (FR), Week 1) will remain on ruxolitinib and dexamethasone. As long as patients show a CR or partial response (PR) at Week 2 (SD15), ruxolitinib and dexamethasone are tolerated, and patients are clinically stable, they will remain on both agents for the remainder of the 8-week study period. Dexamethasone will be weaned every 2 weeks as tolerated. In case of disease reactivation, therapy will be re-intensified.

Patients whose HLH responds unfavorably after 1 week (SD8) of therapy (e.g., unfavorable response, Week 1) will have etoposide added (150 mg/m^2/dose, IV weekly). If patient meets CR or PR at Week 2 (SD15), then combination treatment with ruxolitinib, dexamethasone, and etoposide will be continued until Week 4 disease evaluation (SD 29). If patients have a CR or PR at the Week 4 disease evaluation (SD 29) or later, further etoposide doses may be held at site PI discretion. Dexamethasone weaning may continue beyond the 8-week study period. Patients whose HLH does not respond favorably (e.g., exhibit non-response (NR), progressive disease (PD)) despite treatment with ruxolitinib, dexamethasone, and etoposide will be taken off treatment and salvage therapy will be considered and decided by the treating physician.

Salvage Arm: Patients with relapsed/refractory HLH will be treated on the Salvage Arm. They will not be included in the Safety Phase but will use the same response-adapted approach. Patients may be enrolled on the Salvage Arm as the Safety Phase is ongoing. Patients will receive ruxolitinib 25 mg/m^2/dose by mouth BID and dexamethasone 5 mg/m^2/dose by mouth or IV BID. The first dose of dexamethasone will be given at least 8 hours after the first dose of ruxolitinib for PK testing purposes, but patients will not be excluded if dexamethasone has already been started before starting ruxolitinib. Disease response evaluations will be completed at 1, 2, 4, 6, and 8 weeks. Treatment will be individualized based on response as described for the Expansion Phase of the Frontline Arm. When the MTD of ruxolitinib has been determined on the Safety Phase of the Frontline Arm, it will be the dose used for any additional patients enrolled on the Salvage Arm. Any patients already on the Salvage Arm who show no adverse effects or toxicity at an assigned dose of 25 mg/m^2 BID will be continued on this dose for the 8 week study period.

HLH Reactivation: For patients who initially respond favorably but then worsen (e.g., "reactivate") during the later phases of induction when dexamethasone is weaned, dexamethasone will be increased back to 5 mg/m^2/dose PO/IV BID (10 mg/m^2/day). If the patient is on a reduced dose of ruxolitinib due to prior toxicity(ies), the ruxolitinib dose may be increased to patient's starting dose, provided the prior toxicity(ies) has resolved for at least 1 week. Patients whose HLH responds favorably will continue to receive ruxolitinib and dexamethasone or ruxolitinib, dexamethasone and etoposide. Patients receiving ruxolitinib, dexamethasone and etoposide whose HLH responds unfavorably will be taken off treatment and be considered for an alternative salvage therapy. For patients receiving ruxolitinib and dexamethasone whose HLH responds unfavorably, etoposide may be added. If the response is favorable, the patient will continue on all 3 medications. If the response is unfavorable after adding etoposide, the patient will be taken off treatment and will be considered for an alternative salvage therapy.

All patients with CNS disease will receive intrathecal (IT) MTX and hydrocortisone (HC), per age-based dosing, once per week for up to 4 weeks.

Patients will be followed for one year after starting protocol therapy or 1 year after HSCT (for those undergoing HSCT).

ELIGIBILITY:
Inclusion Criteria: Frontline Arm:

1. Patient is ≥6 weeks and ≤22 years of age.
2. Patient weighs ≥3 kg.
3. Patient is able to take medication PO and/or patient or parent is willing to have NG tube placed if patient is unable to take medications PO.
4. Patient has active HLH if:

   * Patient has ≥5 of 8 Diagnostic HLH criteria listed below, OR
   * Patient has known fHLH (e.g., patient has pathogenic/likely pathogenic germline variant(s) in genes such as PRF1, UNC13D, STX11, STXBP2, LYST, RAB27A, XIAP, SH2D1A, NLCR4) and meets ≥4 of the diagnostic HLH criteria listed below, OR
   * Patient has high likelihood of fHLH based on absent perforin, SAP, XIAP expression and meets ≥4 of the Diagnostic HLH Criteria listed below:

     * Fever
     * Splenomegaly (If present at any point prior to starting study drug)
     * Cytopenias affecting ≥2 of 3 cell lineages in the peripheral blood (hemoglobin <9 g/dL, platelets <100 × 10^9/L, ANC <1000/mm^3)
     * Hypertriglyceridemia (fasting triglycerides ≥265 mg/dL) or hypofibrinogenemia (fibrinogen ≤150 mg/dL)
     * Presence of hemophagocytosis in BM or other tissues
     * Low or absent NK-cell activity (if present at any point prior to starting study drug) OR decreased CD107a mobilization (if present at any point prior to starting study drug)
     * Ferritin ≥500 ng/mL
     * Soluble IL-2 receptor (CD25) ≥2400 U/mL
5. Patient has not received prior HLH therapy, except steroids (any dose or length of therapy is allowed) OR anakinra (any dose or length of therapy is allowed).
6. Patient, parent, or legal authorized representative (LAR) must provide informed consent.

Inclusion Criteria: Salvage Arm:

1. Patient is ≥6 weeks and ≤22 years of age.
2. Patient weighs ≥3 kg.
3. Patient or parent is willing to have the NG tube placed if patient is unable to take medications PO.
4. Patient has past history of HLH, defined as meeting ≥5 of 8 HLH- 2004 diagnostic criteria for those with no known HLH-associated mutations, OR ≥4 of 8 HLH-2004 diagnostic criteria for those with known familial disease.
5. Patient must have active HLH at the time of eligibility assessment, defined as 3 or more of the following Relapsed/Refractory HLH Criteria:

   * Fever
   * Splenomegaly (recurrent or worsening)
   * ANC <1000/mm^3 × 2 assessments over at least 3 days OR platelets <100 × 10^9/L × 2 assessments over at least 3 days, OR need for platelet transfusions
   * Hypofibrinogenemia (fibrinogen ≤150 mg/dL)
   * Soluble IL-2 receptor level ≥ 2400 U/mL
   * Worsening CNS symptoms OR new abnormal brain magnetic resonance imaging (MRI) findings deemed consistent with CNS HLH by the primary treating physician OR CSF cell count ≥5 mm^3 (with or without hemophagocytosis) OR CSF protein higher than the institutional upper limit of normal OR CSF neopterin higher than the institutional upper limit of normal
   * Presence of hemophagocytosis in the BM or other tissues
   * Increasing ferritin × 2 assessments over at least 3 days (both levels must be ≥2000 ng/mL)
6. Patient must be deemed by the primary treating physician to have not responded to prior therapy by either not having or maintaining a response
7. Patient must have received prior HLH-directed therapy:

   * At least 2 weeks of steroids (equivalent to at least 5 mg/m^2/day dexamethasone or 1 mg/kg/day methylprednisolone) AND at least 2 doses of etoposide; OR
   * At least 1 dose of ATG
8. Patient or parent/LAR must provide informed consent.

Laboratory findings must be given on at least 2 assessments, each completed at least 1 day apart, EXCEPT CNS radiologic/laboratory findings in which a single abnormal value is sufficient.

Exclusion Criteria: Frontline and Salvage Arms:

1. Patient is <6 weeks or >22 years of age.
2. Patient weighs <3 kg.
3. Patient has isolated CNS disease.
4. Life expectancy is <2 weeks.
5. Patient is likely to require <4 weeks of therapy (i.e., HSCT is imminent).
6. Patients with creatinine clearance (CrCl) <15 mL/min who are NOT receiving dialysis.
7. Patient has evidence of severe organ dysfunction, defined as: Severe liver dysfunction (ALT >1000 U/L), OR Cardiorespiratory failure requiring any ionotropic support OR extracorporeal life support, OR high frequency oscillatory ventilation, other forms of respiratory support or ventilation are allowed if the patient is not on vasopressors)
8. Patient with pre-existing rheumatologic disorder.
9. Patient with known active malignancy.
10. Patient with previous HSCT, except when HSCT was for treatment of HLH.
11. Patient is pregnant or lactating.
12. Patients who expect to conceive or father children within the projected duration of the study and/or who are unwilling to use highly effective methods of contraception throughout the duration of the study, starting with the screening visit through the end of the treatment visit.
13. Patient has suspected or known fungal disease.
14. Patient is unable to tolerate administration of drugs PO or NG.
15. Patient is taking rifampin or St. John's Wort.
16. Patient is taking another investigational agent or is enrolled on another treatment protocol.
17. Patient, parent, or LAR are unable or unwilling to provide informed consent.

Additional Exclusion Criteria for the Frontline Arm:

1. Patient has or is receiving treatment with a JAK inhibitor (including ruxolitinib), ATG, alemtuzumab, etoposide, tocilizumab, emapalumab or any other HLH-directed therapy other than steroids or anakinra (as defined in the Frontline Arm Inclusion Criteria, #5).

Additional Exclusion Criteria for the Salvage Arm:

1. Patient has or is receiving treatment with a JAK inhibitor (including ruxolitinib) or alemtuzumab within the last 3 months.
2. Patient has received therapy on the Frontline Arm of this trial.

Ages: 6 Weeks to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR)/Complete Response with Incomplete Hematologic Recovery (CRi) | 8 weeks
  Will be reported as number and percentage of patients meeting CR/CRi criteria at the end of 8 weeks of therapy
Adverse events (AEs) associated with the ruxolitinib-containing regimen | up to 8 weeks
  Cumulative incidence will be estimated by the Kalbfleisch-Prentice method for severe toxicities that lead to morbidity and mortality.
Adverse events (AEs) associated with the ruxolitinib-containing regimen | up to 1 year after diagnosis
  Cumulative incidence will be estimated by the Kalbfleisch-Prentice method for severe toxicities that lead to morbidity and mortality.

SECONDARY OUTCOMES:
Overall Response (CR/CRi plus Partial Response [PR])) | 8 weeks
  Will be reported as number and percentage/proportion of patients meeting response (CR/CRi plus PR) criteria at the end of 8 weeks of therapy
Survival to eight weeks | 8 weeks
  The proportion (probability) of patients surviving to the end of 8 weeks will be estimated by sample proportions along with the 95% exact binomial CIs in the Frontline and Salvage Arms, respectively.
Survival to allogeneic hematopoietic stem cell transplantation (HSCT) in patients for whom an allogeneic HSCT is planned | up to 1 year
  The proportion (probability) of surviving to HSCT will be estimated by sample proportions along with 95% exact binomial CIs in the Frontline and Salvage Arms, respectively.
Survival to one year after initiation of the treatment protocol | 1 year after initiation of treatment
  One-year Overall Survival (OS) rate will be estimated in all patients
Survival one year after HSCT | 1 year post HSCT
  One-year post-HSCT Overall Survival (OS) rate will be estimated in patients who receive transplantation, in the Frontline and Salvage Arms, respectively.
Time to Response (CR/CRi or PR) | At weeks 2, 4, 6, and 8
  The mean time to CR/PR including CRi for week 8 response evaluation (will be estimated by the sample mean along with 95% CIs, in the Frontline and Salvage Arms, respectively. The median time will be estimated by the sample median along with the 95% finite- sample CI.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Hines, MD, Study Chair — St. Jude Children's Research Hospital; Kim E. Nichols, MD, Study Chair — St. Jude Children's Research Hospital
Locations (13):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Orange County, Orange, California
  - University of California San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - John Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Children's Wisconsin/Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols